CLINICAL TRIAL: NCT03014284
Title: Novel Listeria Vectors Secreting Gut Flora-Altering Agents to Prevent Colon Cancer and Treat Colitis
Status: Withdrawn | Type: Observational
Why Stopped: Military collaborator sample supplier was transferred, no samples obtained
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS 16-0101; HSC20160555H (Other: UTHSCSA IRB)
Record Dates: First submitted 2016-12-20; First posted 2017-01-09 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-02

CONDITIONS: Colon Cancer; Colitis
Keywords: Tissue collection; colonoscopic surgical procedures
MeSH Terms: conditions — Colonic Neoplasms; Colitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Obtain human colon tissue for ex vivo studies of B7-H1 expression, signaling pathways and effects of recombinant Listeria vectors.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a simple tissue collection study with no therapeutic intent. Colon tissues will be taken from standard of care procedures. Tissues will be tested for their functions, expression of immune co-signaling molecules and reactions to transduction with recombinant Listeria vectors to assess effects on expression of B7-H1 and cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent (or have consent provided through a guardian)
* No immune-modulating drug use during study or within 30 days prior to enrollment
* Having colon material collected as part of standard of care

Exclusion Criteria:

* Unable to provide informed consent (or have consent provided through a guardian)
* Not having colon material collected as part of standard of care

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 50% of patients are expected to be Caucasian, about 40% Hispanic and the remainder African American and other minorities. The investigators anticipate that subjects will range in age from 18 years old and older.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Expression of B7-H1 | Baseline tissue collection
  To assess the ability of recombinant Listeria to modulate B7-H1 in human colonic tissues

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Curiel, MD, Principal Investigator — University of Texas Health Science Center at the Cancer Therapy and Research Center
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States